CLINICAL TRIAL: NCT03977311
Title: A Pilot Study Evaluating the Safety and Feasibility of MR-Guided High-Intensity Focused Ultrasound in Conjunction With Radiation Therapy for the Treatment of Locally Advanced Cervical Cancer
Brief Title: MR-Guided High-Intensity Focused Ultrasound in Conjunction With Radiation Therapy for the Treatment of Locally Advanced Cervical Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to go forward with study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-x066
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MR-HIFU (Experimental): -The study team will determine the tumor volume to be treated per standard-of-care diagnostic MRI or CT imaging. An array of scans will be used to align the participant with the HIFU system, optimize heat delivery to the patients, and/or monitor aspects related to the participant such as motion. Vendor-provided software will be used with the participant in each position to create a customized treatment plan for heat delivery. The HIFU device will then be used to apply clinical levels (41-42°C) of heat to the tumor volume. Regions will be heated to the 41-42°C for up to 60 minutes in one session (either before or after radiation) on one day per five to ten standard radiation therapy fractions, with a maximum of 6 days of hyperthermia over the course of their standard, indicated radiation therapy treatment.
  Interventions: Device: Sonalleve Magnetic Resonance-guided High Intensity Focused Ultrasound (MR-HIFU); Radiation: Radiation therapy

INTERVENTIONS:
Device: Sonalleve Magnetic Resonance-guided High Intensity Focused Ultrasound (MR-HIFU) — -To be used in conjunction with radiation therapy in the treatment of locally advanced cervical carcinoma patients
Radiation: Radiation therapy — -Standard of Care

SUMMARY:
In this study, safety and feasibility of MR-guided HIFU hyperthermia application will be assessed in patients diagnosed with locally advanced cervical cancer. This site has reasonable soft tissue pathways and depths for the ultrasound to access with limited osseous or air interference. Additionally, of cervical cancer patients who develop recurrence following standard treatment, approximately 1/3 will recur locally and an additional 1/3 recur both locally and distantly. Risk of local failure increases with higher FIGO staging. Therefore, patients with locally advanced cervical cancer stand to benefit from adjuvant hyperthermia to potentially increase local disease control outcomes. While MR-HIFU may conceivably increase risk for local complications such as fistula formation, these risks are felt to be acceptable given the potential morbidity of local disease failure, which often can only be addressed curatively by pelvic exenteration. In this study, testing will be performed within tumor volumes involving the cervix uteri. Heating will be to the therapeutic level of 41-42°C for 30-60 minutes, a commonly utilized therapeutic target. This session duration will be achieved in either a single session either before or after the radiotherapy fraction or in an optional two sessions of 15-30 minutes both before and after the radiotherapy fraction, for a total time of 30-60 minutes one day per week. This study will help to elucidate the feasibility of achieving and maintaining therapeutic hyperthermia within an entire tumor volume over the goal period of time of 30-60 minutes.

The investigators anticipate that successful completion of this study will lead to further clinical trials investigating the treatment efficacy in terms of added local control compared to traditional, standard-of-care radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically or cytologically confirmed locally advanced cervical cancer, FIGO Stage IB2 to IVA
* Measurable disease per RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 3 (Karnofsky ≥ 60%)
* Planned treatment includes radiation therapy.
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Currently receiving any investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Pacemaker or other implantable device subject to radiofrequency interference in the ultrasound field.
* Claustrophobia or other contraindications for MRI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MR-HIFU hyperthermia: number of participants who achieve a temperature at or above 41 degrees Celsius | Completion of all participants with their radiation treatment (estimated to be 38 months)
  -Measured by the number of participants who achieve a temperature at or above 41 degrees Celsius within the target region for 2/3 of the intended heating duration in at least 1 MR-HIFU hyperthermia session in at least 5/10 enrolled patients
Number of device/treatment related adverse events recorded by frequency and severity | Through 12 months following completion of treatment (estimated to be 14 months)
  -Severity of adverse events per patient will be evaluated and reported in accordance with the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 standard published by the National Cancer Institute (NCI)

SECONDARY OUTCOMES:
Local control rate | Through 12 months after completion of treatment (estimated to be 14 months)
  -Fraction of patients who remain free of disease in the pelvis following treatment
Comparison of Quality of life as measured by EORTC-QLQ-C30 | Pre-treatment, 3 months after completion of radiation, and 6 months after completion of radiation
  -30 questions about health with 1 = not at all and 4 = very much
  -. Estimate the average of the items that contribute to the scale; this is the raw score then use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score indicates a "worse" level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu